CLINICAL TRIAL: NCT00352833
Title: Multicenter, Open-Label and Randomized Phase II Study to Evaluate Safety and Efficacy of the Trifunctional Bispecific Antibody Catumaxomab (Anti-EpCAM x Anti-CD3) in Patients After Curative Resection of a Confirmed Gastric Adenocarcinoma Compared With Surgery Alone
Brief Title: Safety and Efficacy Study With Catumaxomab in Patients After Curative Resection of a Gastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neovii Biotech (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-REM-GC-02
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2007-10-26 (Estimated); Status verified 2007-06

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma
Keywords: gastric cancer; investigational drug; adjuvant therapy; intraoperative; intraperitoneal; EpCAM-positive tumor
MeSH Terms: conditions — Stomach Neoplasms | interventions — catumaxomab

INTERVENTIONS:
Drug: catumaxomab

SUMMARY:
Investigation of the outcome of an adjuvant treatment with catumaxomab as compared to surgery alone in patients after curative resection of a gastric adenocarcinoma in order to gain more detailed information primary on safety, tolerability and feasibility and secondary on relevant efficacy parameters.

DETAILED DESCRIPTION:
A controlled, randomized, open-label, multi-center, parallel-group, Phase II study to generate valid hypotheses on safety and efficacy issues in patients with a primary confirmed diagnosis of gastric adenocarcinoma and a high risk of disseminated tumor cells due to serosal infiltration after curative gastrectomy. Eligible patients will be centrally randomized by IVRS during operation to one of the two study groups in an 1:1 ratio: surgery plus catumaxomab or surgery alone.

Treatment with catumaxomab will consist of an initial dose of 10 µg given intraoperatively as an intraperitoneal bolus on day 0 and of four following ascending doses (10-20-50-150 µg) which will be administered as an i.p.-infusion via a provided indwelling catheter on the days 7, 10, 13 and 16, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Patient has a primary diagnosis of a histologically confirmed gastric adenocarcinoma (including GE junction Siewert-Type 2 or 3)
* Intended curative gastrectomy ('en-bloc´-R0-resection considering the standard D2-scheme)
* Serosal infiltration (T3/T4, N+/-, M0) confirmed by immediate section with histopathologic assessment during surgery
* Karnofsky index >= 70
* Negative pregnancy blood test at screening in women with childbearing potential

Exclusion Criteria:

* Presence of distant metastases
* Macroscopic and microscopic residual tumor present after surgery
* State after pancreas resection or thoracotomy
* Exposure to prior cancer therapy or planned adjuvant chemo-or radiotherapy of the current gastric cancer
* Previous treatment with non-humanized mouse or rat monoclonal antibodies
* Known/suspected hypersensitivity to catumaxomab or similar antibodies
* Any cancer disease or any cancer treatments within the last 5 years
* Presence of constant immunosuppressive therapy
* Inadequate renal function (creatinine > 1.5 x ULN)
* Inadequate hepatic function (AST or ALT > 2.5 x ULN or bilirubin >= 1.5 x ULN)
* Platelets < 75000 cells/mm³; absolute neutrophil count < 1500 cells/mm³
* Patient had a bowel obstruction within the last 30 days
* Pregnant or nursing woman, or woman of childbearing potential who is not using an effective contraceptive method during the study and at least contraceptives, intrauterine devices, double-barrier method, contraceptive patch, male partner sterilization or condoms)
* Presence of any acute or chronic systemic infection
* Any further condition which according to the investigator results in an undue risk to the patient during participating in the present study
* Patient is an employee of any involved study investigator or any involved institution including the study sponsor
* Parallel participation in another clinical trial or previous participation in this study
* Treatment with another investigational product during this study or during the last 30 days prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
safety and efficacy data

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Heiss, Prof. Dr., Principal Investigator — Cologne, Germany
Locations (1):
- Hospital of Cologne-Merheim, Surgical Department, Cologne, Germany

REFERENCES:
- [Background] Heiss MM, Strohlein MA, Jager M, Kimmig R, Burges A, Schoberth A, Jauch KW, Schildberg FW, Lindhofer H. Immunotherapy of malignant ascites with trifunctional antibodies. Int J Cancer. 2005 Nov 10;117(3):435-43. doi: 10.1002/ijc.21165. PMID 15906359
- [Background] Ruf P, Lindhofer H. Induction of a long-lasting antitumor immunity by a trifunctional bispecific antibody. Blood. 2001 Oct 15;98(8):2526-34. doi: 10.1182/blood.v98.8.2526. PMID 11588051
- [Background] Riesenberg R, Buchner A, Pohla H, Lindhofer H. Lysis of prostate carcinoma cells by trifunctional bispecific antibodies (alpha EpCAM x alpha CD3). J Histochem Cytochem. 2001 Jul;49(7):911-7. doi: 10.1177/002215540104900711. PMID 11410615
- [Background] Zeidler R, Mysliwietz J, Csanady M, Walz A, Ziegler I, Schmitt B, Wollenberg B, Lindhofer H. The Fc-region of a new class of intact bispecific antibody mediates activation of accessory cells and NK cells and induces direct phagocytosis of tumour cells. Br J Cancer. 2000 Jul;83(2):261-6. doi: 10.1054/bjoc.2000.1237. PMID 10901380
- [Background] Zeidler R, Reisbach G, Wollenberg B, Lang S, Chaubal S, Schmitt B, Lindhofer H. Simultaneous activation of T cells and accessory cells by a new class of intact bispecific antibody results in efficient tumor cell killing. J Immunol. 1999 Aug 1;163(3):1246-52. PMID 10415020